CLINICAL TRIAL: NCT05925478
Title: Pterygopalatine Fossa Block in Aneurysmal Subarachnoid Hemorrhage
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Noah Jouett, Fellow Physician, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2023-0176
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental)
  Interventions: Procedure: Ptergyopalatine Fossa Block; Drug: Bupivacaine 0.25% Injectable Solution

INTERVENTIONS:
Procedure: Ptergyopalatine Fossa Block — Injection of local anesthetic (e.g. Bupivacaine) into the pterygopalatine fossa to treat headache related to aneurysmal subarachnoid hemorrhage
Drug: Bupivacaine 0.25% Injectable Solution — Injection of local anesthetic (e.g. Bupivacaine) into the pterygopalatine fossa to treat headache related to aneurysmal subarachnoid hemorrhage

SUMMARY:
Aneurysmal subarachnoid hemorrhage (aSAH) can cause a severe headache (HA) that is famously treatment-resistant. Current pain regimens are too reliant on opioids, which results in long-term opioid dependence and can obfuscate the neurological examination, which is critical to detect vasospasm and delayed cerebral ischemia. This study will gather the initial evidence of whether the pterygopalatine fossa (PPF) regional anesthesia nerve block can treat aSAH-related HA and reduce opioid consumption in patients with aSAH.

ELIGIBILITY:
Inclusion Criteria:

* Aneurysmal subarachnoid hemorrhage with secured aneurysm
* Age greater than or equal to 18 years
* Able to communicate pain level

Exclusion Criteria:

* Documented allergy to local anesthetics (e.g. bupivicaine)
* Patients with unsecured aneurysms
* Patients who are unable to communicate pain level (e.g. sedation/mechanical ventilation/delirium, etc)
* Medical treatment for vasospasm including blood pressure/inotropic augmentation
* Angiographic treatment for vasospasm within 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 3 days
Pain Rating Scale | 3 days
  Scale of 1-10, 1 being lowest possible pain, 10 being highest possible pain

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern, Dallas, Texas, United States